CLINICAL TRIAL: NCT05588895
Title: NOTIFY 2: Picture of Incidental Calcium To Understand Risk Estimate
Brief Title: Picture of Incidental Calcium To Understand Risk Estimate (PICTURE) Trial
Acronym: PICTURE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Fatima Rodriguez, Associate Professor of Medicine (Cardiovascular Medicine), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 67227
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Calcification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Notification (Experimental): The notification arm will have its CT scans interpreted and reported according to standard clinical practice. A standardized notification message using the EHR will be sent to the patient's Stanford affiliated non-EP cardiologist, if present, or the primary care clinician if there is no non-EP cardiologist. After a two week delay from notifying the patient's non-EP cardiologist or PCP, a standardized notification message will be sent to the patient. The message will include an image of the CAC from the chest CT. All communications will be signed by the Principal Investigator. Any treatment decisions will be made by the patient and their clinician.
  Interventions: Other: Notification
- Usual Care (No Intervention): The usual care arm will have its CT scans interpreted and reported according to standard clinical practice. This may mention the presence of CAC in the official radiology imaging report, per usual practice. The usual care arm will not receive any notification beyond this standard of care.
  We intend to notify patients in the usual care arm when study ends, if we determine that notification is effective at increasing statin rates.

INTERVENTIONS:
Other: Notification — For patients randomized to notification, the affiliated non-EP cardiologist, if present, or if patient does not have one, the PCP will be notified and will receive an electronic health record (EHR) message notifying them of the presence of CAC (with images) and the ACC/AHA guideline recommendation to consider starting statin therapy. Simultaneously, the patient will be notified via a MyHealth message describing the presence of CAC with personalized scan images, its significance, and the recommendation that statin therapy should be considered.
  For the notification arm, we will check for either statin prescription or a documented discussion in the EHR at 2 months. For those not prescribed a statin and without a documented discussion in Epic at 2 months follow-up, we will send a repeat notification to their home address and to their affiliated clinician.
  Arms: Notification

SUMMARY:
This is a prospective randomized controlled trial assessing the impact of notifying patients and their clinicians of an incidental finding of coronary artery calcification (CAC) indicating increased cardiovascular risk. Patients will be identified through completed radiology orders for non-gated, non-contrast chest CT in the appropriate clinical context and then will have an EHR screen for inclusion criteria. The presence of CAC will be confirmed by a radiologist. Eligible patients will be randomized to CAC notification or usual care using a 1:1 stratified block randomization method based on baseline ASCVD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above and <85
* Non-gated chest CT with CAC
* An encounter after July 1, 2021 with a Stanford-affiliated clinician from one of the following clinics:

  * Stanford Internal Medicine (includes University affiliated clinics)
  * Stanford Family Medicine (includes University affiliated clinics)
  * Non-EP cardiologist

Exclusion Criteria:

* Advanced or poor-prognostic cancer
* No active primary care or cardiology care at Stanford Health Care
* Primary language other than English, Spanish, Vietnamese, Cantonese, or Mandarin
* Baseline statin or non-statin lipid lowering therapy
* Allergy to statin medication or identification of statin-associated muscle symptom

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of new statin prescriptions | Baseline through Month 6
  6-month new statin prescription rate

SECONDARY OUTCOMES:
Number of participants using statin medication | Month 6
  6-month assessment of statin prescription rates
Change in Low-density lipoprotein (LDL) cholesterol | Baseline and Month 6
Change in 10-Year Atherosclerotic Cardiovascular Disease (ASCVD) Pooled Cohort Equation | Baseline and Month 6
  This outcome measures the 10 year risk of ASCVD events.
Number of events requiring primary care intervention, cardiology referrals, or cardiac testing | Baseline through Month 6
  This outcome assesses healthcare resource use (primary care clinical encounters, cardiology referrals, cardiac testing).

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No